CLINICAL TRIAL: NCT07153536
Title: Spinal Cord Stimulation Combined With Physical Therapy in Post-Stroke Upper-Limb Motor Hemiparesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marco Capogrosso (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Marco Capogrosso, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY25060125; 1UG3NS123135-01A1 (NIH)
Record Dates: First submitted 2025-08-20; First posted 2025-09-04 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Spinal Cord Injuries and Disorders; Hemiparesis After Stroke
Keywords: spinal cord stimulation
MeSH Terms: conditions — Stroke; Spinal Cord Injuries; Disease | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Single-center, interventional, open-label, non-randomized, single-arm feasibility study to obtain initial evidence of safety and efficacy of using spinal cord stimulation (SCS) in combination with physical therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Physical Therapy Alone, then Combined with Spinal Cord Stimulation (Experimental): Two percutaneous leads will be implanted unilaterally on the affected side in the epidural space of the C3-T1 vertebrae (Medtronic Vectris™ SureScan™ 1x8). The leads will be connected to an external stimulator (Medtronic Inceptiv™ spinal cord neurostimulation system) during research activities.
  Interventions: Device: Spinal Cord Stimulator (Medtronic Inceptiv™ System); Other: Physical Therapy

INTERVENTIONS:
Device: Spinal Cord Stimulator (Medtronic Inceptiv™ System) — The Medtronic Inceptiv™ spinal cord neurostimulation system is a rechargeable implantable pulse generator (IPG) designed to deliver electrical pulses to the spinal cord via implanted leads. The system is intended for use in patients with chronic pain.
Other: Physical Therapy — The physical therapy intervention consists of two components: the Mind-Pod Dolphin system (targeting arm function) and the Hummingbird Hunt system (targeting hand function). Both systems use interactive gaming software that enables participants to engage in remote, game-based therapy. Each system offers multiple difficulty levels, allowing participants to progress as their skills improve.

SUMMARY:
This study plans to use systems that have been developed by Medtronic to investigate the use of cervical spinal cord stimulation to treat adults with upper limb hemiparesis resulting from a stroke. The spinal cord stimulation (SCS) will be combined with physical training to improve arm and hand motor control. The study is divided into three phases. In the first phase, after baseline assessments, participants will undergo a Physical Training Protocol (PTP) for 6 weeks including 3 sessions of 90 mins/session per week. After receiving the Medtronic implantable system, in Phase 2, they will then repeat the same PTP program in combination with spinal cord stimulation during the entirety of each of the rehabilitation sessions. Finally, in Phase 3, participants will go home, will not be able to use the stimulation at home but will participate in monthly assessments in the laboratory in which the functionality of the Medtronic system and their motor performances will be assessed for up to 6 months.

DETAILED DESCRIPTION:
The main goal for this study is to evaluate safety of the Medtronic system in the stroke population. The second goal of this study is to assess and document the effects of SCS on motor control. More specifically, whether the combination of SCS and physical exercise (PTP+SCS) will improve motor control and reduce impairments, with the goal of optimizing inclusion criteria and outcome measures for future efficacy studies. To achieve this goal, we designed a study based on the rationale that the ramp up PTP phase 1 will bring people to a plateau motor impairment, in consequence any improvement upon this plateaued level should be due to the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Experienced an ischemic or hemorrhagic stroke that resulted in arm and hand hemiparesis more than 6 months prior to the time of enrollment (Prior strokes that did not cause upper extremity motor deficits are not exclusionary.)
2. Age 22 to 70 years old
3. Upper extremity motor score higher than 20 and lower than or equal to 45 on the Fugl-Meyer Assessment (FMA) scale
4. FMA upper extremity sensory score higher than 6 points (out of 12 points)
5. The ability to communicate, understand, give appropriate consent and follow two-step commands

Exclusion Criteria:

1. Presence of any serious disease or disorder (ex. Neurological conditions other than stroke, cancer, severe cardiac or respiratory disease, renal failure, etc.) that could affect their ability to participate in this study
2. Considered to be at high-risk of recurrent stroke as evident from their medical history or upon judgment of the study physician
3. Presence of post-stroke central pain, other forms of pain or other constraints such as joint contractures in the paretic arm that are serious enough to prevent or affect the correct execution of the physical training protocol as judged by the study therapist
4. A score on the Short Blessed Test assessment scale higher than 9
5. Female participants of child-bearing age who are pregnant or breastfeeding during the study
6. Participants that cannot suspend their antiplatelets and/or anticoagulant therapy for two weeks around the time of surgery
7. Existence of any implanted medical device that is not MRI safe and/or any active medical devices even if it is MRI safe
8. Implanted spinal fusion and stabilization devices such as plates and rods between the C2 and T3 spinal vertebra
9. Obstructed or restricted epidural spinal canal to the point of hindering or increasing the risk of implant of the spinal leads as judged by the study surgeon upon screening imaging
10. Severe claustrophobia that prevents execution of the required MRI imaging sessions
11. Taking anti-spasticity or anti-epileptic medications
12. T-score higher than 63 on the 18-question Brief Symptoms Inventory (BSI-18) who have undergone discussions with and been deemed unsuitable by the Principal Investigator and a study physician

Potential participants who may be excluded on initial screening may discuss possible medication changes with their physician.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number and Severity of Adverse Events | From enrollment to the end of treatment at 49 weeks
  Success Criteria: no serious adverse events related to the stimulation or intolerable. adverse events reported

SECONDARY OUTCOMES:
Motor Impairment - Post Implant to end of Phase 2 | Post implant to the end of Phase 2 (11 weeks)
  The investigators will measure the change in Fugl Meyer (FM) score from post-implant to the end of Phase 2 with SCS ON. The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment. The upper extremity motor function score ranges from 0 to 66 points. Success criteria: mean change FM across Phase 2 is greater than zero, indicating an additional therapeutic benefit of SCS beyond physical training executed in Phase 1 .
Motor Impairment - Absolute Change | Baseline to the end of Phase 2 (19 weeks)
  The investigators will measure the change in Fugl Meyer (FM) score from the baseline to the end of Phase 2 with SCS OFF. The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment. The upper extremity motor function score ranges from 0 to 66 points. Success criteria: mean change FM across the study period is greater than 5, indicating the average improvement surpasses the minimal clinically meaningful threshold.
Spasticity - Phase 2 | Phase 2 (7 weeks)
  The investigators will quantify spasticity scores using the Modified Ashworth Scale (MAS) which is an assessment that is used to measure the increase in muscle tone. MAS assigns a grade of spasticity from a 0-4 ordinal scale. The grade is assigned by moving a joint/muscle through a high velocity quick stretch.
  The investigators will measure the change in MAS score across phase 2. The test is executed with SCS OFF. Success criteria: mean change MAS across Phase 2 is greater than 0. This would show that SCS is able to reduce spasticity beyond the Phase 1 physical training.
Spasticity - Absolute Change | Baseline to the end of Phase 2 (19 weeks)
  The investigators will quantify spasticity scores using the Modified Ashworth Scale (MAS) which is an assessment that is used to measure the increase in muscle tone. MAS assigns a grade of spasticity from a 0-4 ordinal scale. The grade is assigned by moving a joint/muscle through a high velocity quick stretch.
  The investigators will measure the change in MAS score from the baseline to the end of Phase 2. The test is executed with SCS OFF. Success criteria: mean change MAS across the study is greater or equal than 2 points, indicating that average reduction surpasses the minimal clinically meaningful threshold.
Strength - Phase 2 | Phase 2 (7 weeks)
  The investigators will measure changes in isometric torque produced during maximal voluntary contractions across shoulder, elbow and grip strength with SCS ON and SCS OFF. Success criteria: 75% of the participants have significantly higher maximal torques (or forces) with SCS ON compared to SCS OFF in at least 1 movement of at least 1 joint. (e.g. elbow extension). This will confirm that SCS can immediately improve strength.
Motor Control - Phase 2 and 3 | Phase 2 through Phase 3 (31 weeks)
  The investigators will repeat Fugl Meyer (FM) testing within the same session with SCS OFF and SCS ON. The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. The upper extremity motor function score ranges from 0 to 66 points, with a higher score indicating a better outcome. Success criteria: 75% of the participants have higher FM scores with SCS ON compared to SCS OFF of at least 3 points.

CONTACTS AND LOCATIONS:
Overall Officials: George Wittenberg, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, may be shared with other researchers for the purpose of data analysis and collaboration.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available at the end of the trial upon publication of the first manuscript. Estimation is 2 years from enrollment of first participant.
Access Criteria: Data must be directly requested to the PI and will be shared upon completion of necessary data sharing agreement to protect confidential patient information.